CLINICAL TRIAL: NCT05858307
Title: Clinical Application of Serum Anti-Müllerian Hormone (AMH) Measurements
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2022.228
Record Dates: First submitted 2023-02-06; First posted 2023-05-15 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Anti-Müllerian Hormone; Polycystic Ovarian Syndrome; Premature Ovarian Insufficiency; Fertility Issues
Keywords: Anti-Müllerian hormone; Polycystic Ovarian Syndrome; Premature Ovarian Insufficiency; Assisted Reproductive Technology treatment; Predictive value; Reproductive outcomes; AMH; PCOS; POI
MeSH Terms: conditions — Polycystic Ovary Syndrome; Primary Ovarian Insufficiency; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to assess the association of Anti-Müllerian hormone (AMH) with polycystic ovarian syndrome, premature ovarian insufficiency and fertility. The main objectives include the following:

1. To study the level of serum AMH in women with PCOS and to evaluate the utility of serum AMH in the diagnosis of PCOS.
2. To evaluate the level of serum AMH in women with POI and to evaluate the utility of serum AMH in the management of POI.
3. To evaluate the associations of basal AMH level with FSH level and AFC respectively for women undergoing ART treatment.
4. To determine the optimal regimen of gonadotropin for ovarian stimulation for women undergoing ART treatment.
5. To evaluate the predictive value of serum AMH in reproductive outcomes including oocyte quality, embryo quality, pregnancy loss, clinical pregnancy and live birth rate in women undergoing ART treatment.

DETAILED DESCRIPTION:
[Background] Anti-Müllerian hormone (AMH), which level can be assessed in serum, is a product of follicular granulosa cells of preantral and small antral follicles in the ovary. AMH expression increases prior to follicle-stimulating hormone (FSH)-dependent selection (follicles up to 8 mm) and rapidly decreases thereafter (follicles > 8 mm. Thus, serum AMH level is a reliable marker of functional ovarian reserve as it reflects the pool of growing follicles. Since AMH is relatively cycle independent and has no inter-rater variability, it is considered to be a more reliable biomarker of ovarian function across an array of clinical conditions when compared with follicle-stimulating hormone (FSH) and antral follicular count (AFC).

<Association between AMH and polycystic ovarian syndrome (PCOS)> PCOS is a common endocrine disorder that causes menstrual irregularity and hyperandrogenism in women. It affects approximately 4-20% of women of reproductive age. Women with PCOS have been shown to have elevated AMH levels when compared with women without PCOS as there is an increased number of ovarian follicles in PCOS. Therefore, AMH is being increasingly recognised as a marker for the diagnosis of PCOS. However, a specific cutoff value is yet to be determined. When the issue is addressed, serum AMH levels could potentially replace ultrasound in the diagnosis of PCOS as ultrasound is more costly and less accessible.

<Association between AMH and premature ovarian insufficiency (POI)> POI is defined as the cessation of ovarian function before the age of 40 years. Timely diagnosis is important in order to appropriately counsel and treat the patients with POI.

Prompt initiation of hormone replacement therapy is vital to minimise the risk of long-term health complications including osteoporosis and premature cardiovascular disease. AMH levels were significantly low to undetectable in women with POI. Since AMH is independent of the timing in a menstrual cycle, the measurement may be beneficial in the phase of menstrual irregularity and could potentially help to assess the progression of ovarian senescence.

<Associations between AMH and Fertility> Serum AMH level is an important indicator of women's ovarian reserve and a crucial tool in assisted reproductive technology (ART) for the evaluation of women's fertility. A recent systematic review concluded that basal serum AMH is a strong pretreatment predictor of poor response to controlled ovarian stimulation (COS) and correlates with the risk of ovarian hyperstimulation syndrome. As such, clinicians can individualise the stimulation protocols to optimise the ovarian response. In addition, AMH-based prognostication counselling can be provided to patients with realistic expectation regarding the ART outcomes.

Ovarian reserve has a well-established positive correlation with pregnancy outcome. However, current evidence of AMH in the prediction of reproductive outcome following ART treatment remains controversial. Therefore, there is a need to study the predictive value of AMH on pregnancy outcome in women undergoing ART.

[Hypothesis]

1. Serum AMH level is elevated in women with PCOS.
2. Serum AMH level is very low or undetectable in women with POI.
3. Serum AMH level has a significant correlation with FSH and AFC in women undergoing ART treatment.
4. Serum AMH level can predict reproductive outcomes following ART treatment.

[Study design] This is a prospective observational study.

[Methods] Investigators will collect data from patients who undergo management for PCOS and POI in the Department of Obstetrics and Gynaecology at the Prince of Wales Hospital from 2022 to 2026. For patients undergoing investigation of PCOS and POI, routine venous blood tests for AMH and hormonal profile including FSH, luteinizing hormonal (LH), oestradiol (E2) levels will be obtained. For patients undergoing ART treatment, routine venous blood tests for AMH and hormonal profile, and transvaginal ultrasound for AFC will be arranged to assess the patients' ovarian reserve prior to the commencement of treatment. Patients will be recruited and consent will be obtained for the storage of any remaining serum from the blood tests. The stored blood samples will then be retrieved for this study.

[Data processing and analysis] Data analysis will be performed using the Statistical Packages of Social Sciences for Windows (SPSS, Inc). Data will be presented by percentage, mean and standard deviation, and median where appropriate. Comparisons between groups will be carried out by Student T test/Mann-Whitney U test for continuous variables and Chi-square/Fisher's exact test for categorical data. Two-tailed P<0.05 will be considered significant.

[Sample size] All patients fulfilling the inclusion criteria attending the Department of Obstetrics and Gynaecology at the Prince of Wales Hospital from 2022 to 2026 will be recruited. The sociodemographic records of the participants including their menstrual history, routine hormonal results, ovarian reserve assessment and ultrasound assessment of AFC will be obtained. Metabolic screening results and ART treatment records and subsequent laboratory and reproductive outcome will be obtained if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Women attending the Paediatric and Adolescent Gynaecological Clinic and Gynaecological Endocrine Clinic of in the Department of Obstetrics and Gynaecology at the Prince of Wales Hospital for the management of PCOS and POI
* Women attending the Assisted Reproductive Technology (ART) Unit of The Chinese University of Hong Kong for ART treatment

Exclusion Criteria:

* Women with age <10 or ≥45
* Current or past diseases affecting gonadotropin, sex steroid secretion, clearance and excretion

Ages: 10 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The following clients will be included in our study population.
  * Women attending the Paediatric and Adolescent Gynaecological Clinic and Gynaecological Endocrine Clinic of in the Department of Obstetrics and Gynaecology at the Prince of Wales Hospital for the management of PCOS and POI
  * Women attending the Assisted Reproductive Technology (ART) Unit of The Chinese University of Hong Kong for ART treatment
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum anti-Müllerian hormone (AMH) (pmol/L) | Within 1 to 2 months after the day of recruitment
  To evaluate the serum AMH level of women who undergo investigation for polycystic ovarian syndrome (PCOS), premature ovarian insufficiency (POI) or subfertility

SECONDARY OUTCOMES:
Type of gonadotropin used for ovarian stimulation | From the first 1 day to last 1 day of ovarian stimulation during ART treatment
  To assess the type of gonadotropin used for ovarian stimulation for women undergoing ART treatment
Total gonadotropin dose used for ovarian stimulation | On the last 1 day of ovarian stimulation during ART treatment
  To assess the total gonadotropin dose used for ovarian stimulation for women undergoing ART treatment
Number of oocytes retrieved | On the 1 day of oocyte retrieval during ART treatment
  To evaluate the number of oocytes retrieved during oocyte retrieval for women undergoing ART treatment
Serum follicle stimulation hormone (FSH) (IU/L) | On the first 1 day of ovarian stimulation during ART treatment
  To evaluate the serum FSH level of women who undergo ART treatment
Serum luteinising hormone (LH) (IU/L) | On the first 1 day of ovarian stimulation during ART treatment
  To evaluate the serum LH level of women who undergo ART treatment
Serum estradiol (pmol/L) | On the first 1 day of ovarian stimulation during ART treatment
  To evaluate the serum estradiol level of women who undergo ART treatment
Antral follicle count (AFC) | On the first 1 to 4 days of ovarian stimulation during ART treatment
  To evaluate the AFC of women who undergo ART treatment
Clinical pregnancy rate | 6 to 7 weeks of gestation
  To assess for the presence of gestational sac using ultrasonography after embryo transfer procedure for women undergoing ART treatment
Live birth rate | from 24 weeks of gestation up to 40 weeks
  To assess whether live babies are born after women receive ART treatment

CONTACTS AND LOCATIONS:
Overall Officials: PUI WAH JACQUELINE CHUNG, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong